CLINICAL TRIAL: NCT02836912
Title: The Efficacy of Pulmonary Rehabilitation Exercise in Home Care for the Non-invasive Ventilator-dependent Elderly With Chronic Obstructive Pulmonary Disease
Brief Title: The Efficacy of Pulmonary Rehabilitation Exercise in Home Care for the Non-invasive Ventilator-dependent Elderly With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-E(I)-20150203
Record Dates: First submitted 2016-07-01; First posted 2016-07-19 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Pulmonary Disease
Keywords: Rehabilitation
MeSH Terms: conditions — Lung Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regular education (No Intervention): Regular education for COPD, including percussion and posture drainage.
- Exercise (Experimental): Besides the same information for the education group, exercise of upper extremity without loading, exercise of lower extremity, and training of respiratory muscles are used for the exercise group.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Besides the same information for the education group, exercise of upper extremity without loading, exercise of lower extremity, and training of respiratory muscles are used for the exercise group
  Arms: Exercise

SUMMARY:
Pulmonary rehabilitation exercise is beneficial for individuals with chronic obstructive pulmonary disease (COPD). However, merely 30% patients know how to do the exercise correctly. Therefore, it is worthy to investigate the applications in clinical practice. In addition, there are no relative research in Taiwan to see effects of an 8-week pulmonary rehabilitation exercise in home care for the non-invasive ventilator-dependent elderly with COPD.

DETAILED DESCRIPTION:
According to estimation of the world health organization (WHO), chronic obstructive pulmonary disease (COPD) would become the third major cause of death. Moreover, the lung recovery exercise is proven beneficial for mild, moderate, or severe COPD by the guideline of GOLD. However, research in Taiwan focused on follow-up medical status for mild or moderate COPD in clinics, or weaning of severe COPD in intensive care unit (ICU). There was no relative research investigating non-invasive ventilator-dependent elderly with COPD on home care. Therefore, this study would explore effects of pulmonary rehabilitation exercise for this group. The pulmonary rehabilitation exercise program in this study is divided into two stages in the experimental group. The first four weeks, 10 minutes for each training (upper extremity without loading, exercise of lower extremity, and respiratory muscles), and totally 30 minutes is required. Consequent four weeks, 15 minutes for upper extremity without loading, 15 minutes for exercise of lower extremity, and 10 minutes for training of respiratory muscles, and totally 40 minutes is scheduled.

ELIGIBILITY:
Inclusion Criteria:

1. age > 65 y/o, and is diagnosed with COPD;
2. is non-invasive ventilator-dependent in home care;
3. is stable evaluated by a doctor;
4. is conscious clear and can perform the exercise (upper, lower extremity, and respiratory muscle training);
5. do not accept exercise training as (4)-mentioned currently

Exclusion Criteria:

1. conscious is not clear enough to perform the exercise training;
2. cannot leave his/her bed independently;
3. cannot wean a ventilator and need to use for 24 hours;
4. severe heart disease (eg. acute myocardial infarction, severe arrhythmia);
5. Oxygen saturation (SPO2) lower than 90% during oxygen therapy
6. fever or acute infections
7. reject to sign consent form
8. age < 20 y/o

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2016-07-26 (Actual); Study Completion 2016-09-26 (Actual)

PRIMARY OUTCOMES:
changed strength of respiratory muscles | baseline , 8 weeks, 12 weeks
  inspforce(BUEHRINGER.USA)

SECONDARY OUTCOMES:
changed lung function | baseline , 8 weeks, 12 weeks
  spirometry
changed value for quality of life | baseline , 8 weeks, 12 weeks
  ST.George's Respiratory Questionnaire
changed score of intensity of dyspnea | baseline , 8 weeks, 12 weeks
  Borg dyspnoea scale
time of weaning from ventilator | baseline , 8 weeks, 12 weeks
  time of using ventilator data is directed recorded continually by chip of his/her ventilator during the study

CONTACTS AND LOCATIONS:
Overall Officials: Miao-Ju Hsu, PHD, Principal Investigator — 100,Shih-Chuan 1st Road,Kaohsiung,80708,Taiwan

IPD SHARING:
Plan to Share IPD: No